CLINICAL TRIAL: NCT04092556
Title: Exploratory Study to Evaluate the Effective Site for Control of Motor Coordination Function After Transcranial Direct Current Stimulation in Multiple Systemic Atrophy With Cerebellar Feature
Brief Title: tDCS for Multiple System Atrophy With Cerebellar Feature
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jinyoung Youn, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-10-010-002
Record Dates: First submitted 2019-09-08; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Multiple System Atrophy, Cerebellar Variant (Disorder)
Keywords: Multiple System Atrophy; Cerebellar Ataxia; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Multiple System Atrophy; Cerebellar Ataxia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS (M1) (Active Comparator): The participants will be submit to tDCS applied over the motor cortex (M1)
  Interventions: Device: transcranial direct current stimulation
- tDCS (Cerebellar cortex) (Active Comparator): The participants will be submit to tDCS applied over the cerebellar cortex
  Interventions: Device: transcranial direct current stimulation
- Sham stimulation (Sham Comparator): The participants will be submit to sham stimulation
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — tDCS involves application of very low amplitude direct current via surface scalp electrodes. The applied current modifies the transmembrane neuronal potential and thus influences the level of excitability. Depending on the polarity of active electrodes tDCS can increase or decrease the cortical excitability.
  Other Names: tDCS

SUMMARY:
The aim of study is to investigate most effective site for control the motor coordination using transcranial direct current stimulation in multiple system atrophy with cerebellar feature

DETAILED DESCRIPTION:
Participants receive transcranial direct current stimulation (tDCS) over M1, cerebellar cortex or sham stimulation for 30 minutes. The type of stimulation depends on random assignment. The participants have a 1 week of wash out period between each stimulation.

The assessment will be done by International Cooperative Ataxia Rating Scale (ICARS), GAITRITE (CIR Systems Inc., Clifton, New Jersey, USA) and PEDOSCAN (DIERS PEDO, Germany) at baseline and immediately after each treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who meet the clinical criteria for probable multiple system atrophy with cerebellar features (MDS second consensus statement on the diagnosis of multiple system atrophy)
* 2. Patients aged between 40 and 70
* 3. Patients who do not have rigidity and bradykinesia
* 4. Patients who have given voluntary consent after understanding the content of the clinical trial

Exclusion Criteria:

* 1. Patients with a serious cognitive disorder, behavioral disorder, or mental illness
* 2. Patients have history of seizure, stroke, encephalitis, other degenerative neurological disease
* 3. Patients with a serious medical disease

  * Patients who concomitantly suffer from severe renal impairment, convulsions, stomach ulcers, moderate or more severe liver disease
  * Patients with un-controlled high blood pressure or diabetes
* 4. Patients who have taken another investigational products within 4 weeks prior to being enrolled in this clinical trial, or patients who are pregnant or breastfeeding

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change from International Cooperative Ataxia Rating Scale (ICARS) | per session: at baseline and within 30 minutes tDCS treatment completion
  The scale is scored out of 100 with 19 items and 4 subscales of postural and gait disturbances, limb ataxia, dysarthria, and oculomotor disorders. Higher scores indicate higher levels of impairment.

SECONDARY OUTCOMES:
Change from temporospatial parameters of gait | per session: at baseline and within 30 minutes tDCS treatment completion
  Gait parameters measured by GAITRite system
Change from posturography | per session: at baseline and within 30 minutes tDCS treatment completion
  Posturography measured by Pedoscan system

CONTACTS AND LOCATIONS:
Overall Officials: Jinyoung Youn, Principal Investigator — Samsung Medical Center, Department of Neurology
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No